CLINICAL TRIAL: NCT00654992
Title: Prevention of Acute Kidney Injury (AKI) by Erythropoietin (EPO) in Patients Undergoing Coronary Artery Bypass Grafting (CABG) Surgery - A Prospective Placebo-Controlled Randomized Trial
Brief Title: Effect of Erythropoietin (EPO) in Kidney After Cardiac Surgery
Acronym: EPO-CABG
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Ki Young Na/MD PhD, Department of Internal Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SNUBH B-0608/036-004
Record Dates: First submitted 2008-04-04; First posted 2008-04-09 (Estimated); Results first posted 2009-06-16 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-04

CONDITIONS: Kidney Failure, Acute
MeSH Terms: conditions — Acute Kidney Injury | interventions — epoetin beta; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EPO group (Active Comparator)
  Interventions: Drug: Erythropoietin-Beta
- Placebo group (Placebo Comparator)
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Erythropoietin-Beta — 300 IU/kg of EPO or saline intravenously before surgery
  Other Names: recormon
  Arms: EPO group
Drug: Normal Saline — 300 IU/kg of normal saline intravenously before surgery
  Other Names: 0.9% saline
  Arms: Placebo group

SUMMARY:
The purpose of this study is to determine whether erythropoietin is effective in preventing acute kidney dysfunction after coronary artery bypass grafting surgery.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) occurs in 7% to 40% of patients undergoing cardiac surgery, depending on the definition of AKI used. Even small increments in serum creatinine have been shown to be associated with increased mortality after cardiac surgery. However, there are no proven interventions to prevent AKI after cardiac surgery. Erythropoietin (EPO) has been shown to have tissue-protective effects in various experimental models. In this prospective placebo-controlled randomized trial, we evaluated the effectiveness of EPO in the prevention of AKI after coronary artery bypass grafting (CABG).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective CABG over age 18

Exclusion Criteria:

* Under age 18
* Emergent CABG
* Prior exposure to nephrotoxic drug
* Dialysis patients
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2006-09; Primary Completion 2008-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ki Young, Na, MD PhD, Principal Investigator — Department of Internal Medicine
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Nishiwaki H, Abe Y, Suzuki T, Hasegawa T, Levack WM, Noma H, Ota E. Erythropoiesis-stimulating agents for preventing acute kidney injury. Cochrane Database Syst Rev. 2024 Sep 20;9(9):CD014820. doi: 10.1002/14651858.CD014820.pub2. PMID 39301879

RESULTS

PARTICIPANT FLOW:
Groups:
- Erythropoietin (EPO) Group: received 300 U/kg of erythropoietin intraveously following induction of anesthesia
- Placebo Group: received normal saline intraveously following induction of anesthesia
Period: Overall Study
Arm/Group | Erythropoietin (EPO) Group | Placebo Group
Started | 36 | 35
Completed | 36 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erythropoietin (EPO) Group | Placebo Group | Total
Number analyzed (Participants) | 36 | 35 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 15 | 14 | 29.0
  >=65 years | 21 | 21 | 42.0
Age Continuous [Mean (Standard Deviation); unit: years] | 65 (11) | 69 (8) | 67 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 18.0
  Male | 30 | 23 | 53.0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 36 | 35 | 71.0

OUTCOME MEASURES:

1. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (eGFR)
Description: estimated glomerular filtration rate (eGFR)as ml/min/1.73m2
Time Frame: during the first 5 days after surgery
Measure: Mean (Standard Deviation); unit: ml/min/1.73m2
Arm/Group | Erythropoietin (EPO) Group | Placebo Group
Number analyzed (Participants) | 36 | 35
ml/min/1.73m2 | -1.5 (7.3) | -9.1 (14.5)

2. Primary Outcome: Number of Participants Who Had AKI (Acute Kidney Injury)
Description: number of participants who had 50% increase in serum creatinine levels from baseline
Time Frame: at any time within the first 5 days after surgery
Measure: Number; unit: participants
Arm/Group | Erythropoietin (EPO) Group | Placebo Group
Number analyzed (Participants) | 36 | 35
participants | 3 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes